CLINICAL TRIAL: NCT07036120
Title: A Study on the Biomechanical Mechanisms of Orthotic/Physical Training Correction of Hallux Valgus and Its Impact on the Lower Limbs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wan Xinzhu (Other)
Responsible Party: Sponsor-Investigator, Wan Xinzhu, Principal Investigator, Master's Candidate, Department of Basic Medical Sciences, Southern Medical University, Southern Medical University, China
Organization: Southern Medical University, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NFYKX003
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hallux Valgus Deformity
MeSH Terms: interventions — Orthotic Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OR group (Experimental): The orthotic group was asked to wear a prefabricated toe orthotic (FORTH, China) on both feet at night each day, which was uniformly procured through an online shopping route prior to the start of the intervention. Subjects were required to wear the orthotics for a minimum of 8 hours per day and were monitored by uploading photos daily. Before the start of the intervention, the patients were instructed on the use of the orthoses and were given a demonstration of wearing the orthoses.
  Interventions: Device: orthosis
- EX group (Experimental): The exercise training group was asked to implement an exercise program for no less than days 5 days per week, and in addition to the fascia ball and elastic bands (LI-NING, China) required for training, subjects were also given a document containing a textual description of the exercise program and a prerecorded video of the actual exercise, which contained information about the exercise position, number of repetitions, duration of contraction, rest time between sets, frequency, and precautions. They were monitored by uploading daily exercise hours and photos, and problems affecting their compliance were addressed.
  Interventions: Behavioral: foot exercises

INTERVENTIONS:
Device: orthosis — (1) one pair of two orthoses, regardless of the right and left sides; (2) loosen the two Velcro straps, put the large Velcro strap into the arch of the foot, and put the small Velcro strap on the thumb; (3) place the rigid plastic fixation plate along the medial edge of the foot and align the axis of rotation with the 1st metatarsalphalangeal joint; (4) tighten the Velcro straps as much as possible to prevent dislocation of the orthoses, without interfering with sleep; (5) tighten the Velcro straps to prevent dislocation of the orthoses, and to prevent the orthoses from moving out of position. Tighten the Velcro straps as much as possible without disturbing sleep to prevent the orthosis from shifting and to position the phalanx correctly in the outer table. Contact the laboratory staff for a new pair of orthotics if the adhesive tape is not sufficiently sticky to maintain positional fixation during sleep.
  Arms: OR group
Behavioral: foot exercises — 1. Warm-up: 30 seconds per movement
     1. Joint loosening
     2. Plantar relaxation
  2. Toe spreading: 10 reps/set, 3 sets/day
  3. Toe grasping towel: 10 times/set, 3 sets/day
  4. Standing Heel Raise: 10 times/group, 3 groups/day
  5. Short Foot Exercise: 10 times/sets, 3 sets/day
  6. Relax the soles of the feet again at the end of all exercises.
  Arms: EX group

SUMMARY:
The study population of this project is mainly young people. Our goal is to investigate the kinematic and kinetic characterization brought about by different conservative treatment modalities for hallux valgus. The main study involves recruiting volunteers, grouping them into 12-week interventions with orthotics or foot exercises, and analyzing the kinematic and kinetic alterations in young and middle-aged subjects before, during, and after cessation of the interventions by motion capture, surface electromyography, and musculoskeletal ultrasound. A database of human biomechanical characteristics was constructed through in-vivo exercise techniques to analyze changes in the biomechanical characteristics of the population with hallux valgus after the use of different intervention methods.

ELIGIBILITY:
Inclusion Criteria:

* Hallux valgus angle > 15°
* Age 18-45 years
* Right leg dominant (based on the Waterloo Foot Questionnaire)
* Bilateral hallux valgus

Exclusion Criteria:

* History of lower limb surgery or neuromuscular diseases causing gait abnormalities (such as lumbar disc herniation and chronic ankle instability)
* Any treatment for hallux valgus within the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Measuring muscle synergy using a 16-channel surface electromyography device | From baseline to 12 weeks of intervention
  The Pearson correlation coefficient (r) was used to measure the independence of individual modules and the consistency of synergistic effects among individuals in the same group. When r > 0.7, it was considered that there was similarity between the two synergy modules. Muscles with a median value > 0.3 in the spatial components of the module were considered to be activated muscles in that module.
Measuring kinematic synergy using optical infrared cameras | From baseline to 12 weeks of intervention
  The Pearson correlation coefficient (r) was used to measure the independence of individual modules and the consistency of synergistic effects among individuals in the same group. When r > 0.7, it was considered that there was similarity between the two synergy modules. Degree of freedom (DoF) with a median value > 0.25 in the spatial components of the module were considered to be activated DoF in that module.

SECONDARY OUTCOMES:
Measuring hallux valgus angle with a protractor | From baseline to 12 weeks of intervention
  The hallux valgus angle between the longitudinal axis of the 1st metatarsal and the longitudinal axis of the proximal phalanx of the 1st toe was measured using a protractor
Using ultrasound diagnostic system to capture a cross-sectional image of the thickest part of the muscle for measuring the cross-sectional area of the muscle | From baseline to 12 weeks of intervention
  Using SONIMAGE HS1 ultrasound diagnostic system to capture a cross-sectional image of the abductor hallucis, flexor hallucis brevis, and flexor digitorum brevis on the right side in a static position. Repeat image acquisition three times, measure the cross-sectional area using software, and take the maximum value.
Using a force plate to measure the center of foot pressure | From baseline to 12 weeks of intervention
  Foot pressure center (COP) data collected during gait testing is standardized according to the physical characteristics of the test subject to generate COP total trajectory length (COP-D), medial and lateral COP deviation (COP-X), and anterior-posterior COP deviation (COP-Y).

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Y, Liu R, Wan X, Chen C, Wang Y, Yu W, OuYang J, Qian L, Liu G. The Effect of Short-Term Kinesiology Taping on Neuromuscular Controls in Hallux Valgus During Gait: A Study of Muscle and Kinematic Synergy. IEEE Trans Neural Syst Rehabil Eng. 2024;32:3199-3209. doi: 10.1109/TNSRE.2024.3451651. Epub 2024 Sep 5. PMID 39208038